CLINICAL TRIAL: NCT06108791
Title: High vs Low Inspired Intraoperative Oxygen Concentration on the Incidence of Surgical Site Infection in Hepatobiliary Surgeries
Brief Title: Intraoperative Oxygen Concentration on Incidence of Surgical Site Infection
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Shimaa Abbas Hassan, lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SSI32641
Record Dates: First submitted 2023-10-25; First posted 2023-10-31 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Surgical Site Infection
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HIGH FIO2 (Active Comparator): will include 50 patients: each one will receive intraoperatively a high concentration of oxygen (80% oxygen + 20% air), following extubation, high-concentration oxygen supplementation will be maintained and given through non-rebreathing face mask with a reservoir at 10 L/min for 2 h.
  Interventions: Drug: FIO2=0.8
- LOW FIO2 (Placebo Comparator): will include 50 patients: each one will receive intraoperatively standard concentration oxygen (33% oxygen + 66% air) followed by oxygen supplementation through the standard Venturi face mask of 30%
  Interventions: Drug: FIO2=0.33

INTERVENTIONS:
Drug: FIO2=0.8 — the concentration of intraoperative inspired fraction of oxygen is 80% oxygen + 20% air
  Arms: HIGH FIO2
Drug: FIO2=0.33 — the concentration of intraoperative inspired fraction of oxygen is 33% oxygen + 66% air
  Arms: LOW FIO2

SUMMARY:
Surgical site infections (SSI) are the most common healthcare-associated infections and sources of morbidity and over-mortality. Factors that have been proven to reduce SSI include antimicrobial prophylaxis, maintenance of perioperative normothermia, avoidance of hyperglycemia, proper surgical techniques, and adequate pain relief postoperatively

DETAILED DESCRIPTION:
In 2016, a systematic review and meta-analysis assessing the effects of systematic high FiO2 (80%) compared with standard FiO2 (30%) concluded that high FiO2 was associated with a reduction of SSI in patients undergoing surgery under general anesthesia. Consequently, the WHO recommended that "adult patients undergoing general anesthesia should receive an 80% FiO2 intra-operatively to reduce the risk of SSI".These recommendations have sparked a large debate on the benefits and harms of hyperoxemia. From the theoretical point-of-view, several pro (prevention of hypoxemia, SSI, and postoperative nausea and vomiting) and con (respiratory adverse events, increased production of harmful "reactive oxygen species") arguments have been raised by believers and detractors of high FiO2. Accordingly, and despite these recommendations, anesthetists still used a wide range of intraoperative FiO2 in daily practice and frequently changed FiO2 settings during surgery unrelated to patients' PaO2 or SpO2.

The PROXI study, the largest multicenter randomized controlled trial specifically designed to assess the role of high vs. low intraoperative FiO2 on SSI, did not report any reduction of the incidence of SSI with the administration of 80% FiO2 during colorectal surgery. Similarly, the recent multicenter randomized iPROVE-O2 trial that included 740 patients undergoing major abdominal surgery, ventilated intraoperatively with an evidence-based protective strategy, reported a similar SSI rate between the 30% and 80% FiO2 groups.

ELIGIBILITY:
Inclusion Criteria:

* - BMI of <35 kg/m2
* scheduled for elective abdominal laparotomy/ laparoscopy under general anesthesia with an expected surgical time longer than 2 h.
* ASA I and II

Exclusion Criteria:

* - Patients undergoing minor procedures, where the expected duration of surgery will be less than 1 hour.
* emergency surgeries for bowel obstruction.
* abdominal surgery for vascular or plastic indications.
* patients with a recent history of fever,
* patients with uncontrolled diabetes mellitus,
* patient with known immunological dysfunction (on steroids, decompensated liver disease, HIV, etc.).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-04-03 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Incidence of SSI | 30 DAYS
  - the incidence of SSI postoperatively according to the Centers for Disease Control (CDC) criteria up to 30 days

SECONDARY OUTCOMES:
Pulmonary complications | 14 days
  defined as the need for controlled ventilation or arterial oxygen saturation below 90% despite supplemental oxygen.

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol